CLINICAL TRIAL: NCT00427349
Title: A Phase II Clinical and Biologic Study of AMG 706 and Octreotide in Patients With Low-Grade Neuroendocrine Tumors
Brief Title: AMG 706 and Octreotide in Treating Patients With Low-Grade Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000526256; ECOG-E4206 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA023318 (NIH)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Neoplastic Syndrome
Keywords: localized gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; gastrinoma; insulinoma; WDHA syndrome; glucagonoma; pancreatic polypeptide tumor; somatostatinoma; recurrent islet cell carcinoma; neuroendocrine tumor
MeSH Terms: conditions — Adenoma, Islet Cell; Neoplasms; Gastrinoma; Insulinoma; Vipoma; Glucagonoma; Somatostatinoma; Carcinoma, Islet Cell; Neuroendocrine Tumors | interventions — motesanib diphosphate; Octreotide; batifiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMG 706+Octreotide (Experimental): Patients receive oral AMG 706 and octreotide acetate intramuscularly (IM) once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  AMG 706 was administered on a flat scale of mg/day and not by weight or body surface area (BSA). AMG 706 was provided as a 25 mg tablet; the daily dose was 125 mg administered as five 25 mg tablets in the morning. AMG 706 was taken daily without breaks in treatment.
  One dose consisted of octreotide-LAR 30 mg administered IM on day 1 of each cycle. The first octreotide-LAR injection would correspond with the first day of AMG 706 and then on day 1 of subsequent cycles.
  Interventions: Drug: AMG 706; Drug: octreotide

INTERVENTIONS:
Drug: AMG 706 — AMG 706 was administered on a flat scale of mg/day and not by weight or body surface area (BSA). AMG 706 was provided as a 25 mg tablet; the daily dose was 125 mg administered as five 25 mg tablets in the AM. AMG 706 was taken daily without breaks in treatment
  Other Names: motesanib diphosphate
Drug: octreotide — One dose consisted of octreotide-LAR 30 mg administered IM on day 1 of each cycle. The first octreotide-LAR injection would correspond with the first day of AMG 706 and then on day 1 of subsequent cycles.
  Other Names: L-cysteinamide; Sandostatin; SMS 201-995

SUMMARY:
RATIONALE: AMG 706 and octreotide may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well AMG 706 and octreotide work in treating patients with low-grade neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 4-month progression-free survival (PFS) of patients with low-grade neuroendocrine tumors treated with AMG 706 and octreotide acetate.

Secondary

* Determine the response rate and overall survival of patients treated with these drugs.
* Determine the toxicity and tolerability of AMG 706 in these patients.
* Determine the effect of AMG 706 on tumor perfusion by functional computerized tomography (CT) scan.
* Determine the effect of AMG 706 on tumor markers (e.g., chromogranin A, 5-hydroxyindoleacetic acid, and gastrin) specific for neuroendocrine tumors.
* Determine the effect of AMG 706 on serum vascular endothelial growth factor (VEGF) levels.
* Determine the expression of VEGF, VEGF receptor-2 (VEGFR-2), chromogranin A, human achaete-scute homolog-1 (hASH1), and Notch1 markers of neuroendocrine tumors.

OUTLINE: This is a multicenter study.

Patients receive oral AMG 706 and octreotide acetate intramuscularly once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Plasma samples are collected at baseline, periodically during study treatment, and at 4 weeks after the completion of study treatment. Samples are used to determine plasma VEGF levels. Gene expression of downstream markers of Raf kinase expression (raf, MEK, and ERK) as well as hASH1 and Notch1 are evaluated at baseline. Tumor tissue collected at diagnosis or prior surgery is examined by reverse transcriptase-polymerase chain reaction assay. Contrast CT scans are conducted at baseline, day 2 of course 1, and week 8 to assess tumor perfusion.

After the completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed low-grade neuroendocrine neoplasm
* Measurable disease
* Radiographic evidence of disease progression after any prior systemic therapy, chemoembolization, bland embolization, or observation, defined by either of the following:

  * Appearance of a new lesion
  * At least 20% increase in the longest diameter of any previously documented lesion or in the sum of the longest diameters of multiple lesions
* Tissue block from original diagnostic or surgical specimen required
* Concurrent stable-dose octreotide acetate required
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be able to receive a contrast-enhanced CT scan
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin level ≥ 8.0 g/dL
* Bilirubin ≤ 2.0 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 3 times ULN (5 times ULN if liver metastases are present)
* Left Ventricular Ejection Fraction (LVEF) ≥ institutional lower limit of normal as evaluated by echocardiography or multigated acquisition (MUGA) scan
* No history of uncontrolled hypertension (resting blood pressure > 150/90 mm Hg)

  * Antihypertensive medications allowed if patients is stable on their current dose
* One prior systemic chemotherapy regimen for low-grade neuroendocrine neoplasm allowed

  * Chemoembolization is not considered systemic chemotherapy
* At least 4 weeks since prior major surgery, chemotherapy, radiation therapy, other systemic therapy, or local liver therapy

Exclusion criteria:

* Prior procedures that would adversely affect intestinal absorption
* Prior anti-vascular endothelial growth factors
* Concurrent chemotherapy or radiation therapy
* History of the following within the past 12 months:

  * New York Heart Association class III or IV congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction
  * Symptomatic cardiac arrhythmia
  * Cerebrovascular accident or transient ischemic attack
  * Arterial or venous thrombosis
* Known history of allergic reactions to AMG 706 or derivatives or to octreotide acetate injections
* Gastrointestinal tract disease resulting in an inability to take oral medication (i.e., ulcerative disease, uncontrolled nausea, vomiting, or diarrhea, bowel obstruction, or inability to swallow tablets)
* Pregnant or nursing
* Small cell lung cancer, medullary thyroid cancer, paraganglioma, or pheochromocytoma
* Requirement for intravenous alimentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (112):
- United States (112):
  - Hematology Oncology Associates of Illinois - Berwyn, Berwyn, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology & Oncology Care, Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin

REFERENCES:
- [Derived] Lubner S, Feng Y, Mulcahy M, O'Dwyer P, Giang GY, Hinshaw JL, Deming D, Klein L, Teitelbaum U, Payne J, Engstrom P, Stella P, Meropol N, Benson A. E4206: AMG 706 and Octreotide in Patients with Low-Grade Neuroendocrine Tumors. Oncologist. 2018 Sep;23(9):1006-e104. doi: 10.1634/theoncologist.2018-0294. Epub 2018 May 31. PMID 29853660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on September 16, 2008, accrued its first patient on November 7, 2008, and closed on March 18, 2010 with 46 patients registered to the study from 10 ECOG-ACRIN affiliated institutions.
Groups:
- AMG 706+Octreotide: Patients receive oral AMG 706 and octreotide acetate intramuscularly once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  AMG 706: AMG 706 was administered on a flat scale of mg/day and not by weight or body surface area (BSA). AMG 706 was provided as a 25 mg tablet; the daily dose was 125 mg administered as five 25 mg tablets in the AM. AMG 706 was taken daily without breaks in treatment.
  octreotide: One dose consisted of octreotide-LAR 30 mg administered IM on day 1 of each cycle. The first octreotide-LAR injection would correspond with the first day of AMG 706 and then on day 1 of subsequent cycles.
Period: Overall Study
Arm/Group | AMG 706+Octreotide
Started | 46
Eligible | 45
Treated | 45
Eligible and Treated | 44
Completed | 0 (Treatment continued until disease progression or intolerable toxicity)
Not Completed | 46
Not completed — Lack of Efficacy | 23
Not completed — Adverse Event | 14
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Alternative therapy | 1
Not completed — Other | 2
Not completed — Ineligible | 1
Not completed — Never started therapy | 1

BASELINE CHARACTERISTICS:
Population: Per protocol, the primary population for all efficacy analysis is all eligible and treated patients
Arm/Group | AMG 706+Octreotide
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Four-month Progression-free Survival Rate
Description: Four-month progression-free survival (PFS) rate is defined as number of patients who are still progression free at 4 months after study entry divided by number of eligible and treated patients enrolled to the study. Progression is evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s), or unequivocal progression of existing non-target lesions.
Time Frame: assessed every 4 weeks while on treatment and at three months post-treatment for participants treated for one cycle, up to month four
Population: The analysis population includes all 44 eligible and treated patients. But 2 patients did not have disease assessment after study entry and are excluded from the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | AMG 706+Octreotide
Number analyzed (Participants) | 42
percentage of participants | 78.5 [65.6 to 88.3]
Statistical Analysis 1: Comparison: AMG 706+Octreotide; The null hypothesis is that the 4-month progression free survival rate is 20%. Alternatively, AMG 706 will be considered worthy of further study if its true progression-free survival rate is 40% or better at 4 months (alternative hypothesis); Test type: Superiority or Other; p < 0.001, one sample binomial test; The study result was compared to a null hypothesis of 20% 4-month progression free survival rate using one sample binomial test

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from registration until death (event), or censored at last date known alive. OS was estimated using the Kaplan-Meier method , with 95% confidence intervals calculated using Greenwood's formula
Time Frame: assessed every 3 months if patient is < 2 years from study entry, then every 6 months up to 5 years
Population: All eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 706+Octreotide
Number analyzed (Participants) | 44
months | 27.5 [14.6 to 45.1]

3. Secondary Outcome: Objective Response Rate
Description: Tumor response was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Objective response rate is defined as number of patients with complete response (CR) or partial response (PR) divided by the total number of analyzable patients. CR is defined as complete disappearance of all tumor lesions, and partial response is defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: assessed every 8 weeks while on treatment, and frequency of tumor measurements during follow-up were determined by the treating physician, assessed up to 5 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | AMG 706+Octreotide
Number analyzed (Participants) | 44
percentage of participants | 13.6 [6 to 25]

ADVERSE EVENTS:
Time Frame: Assessed at the end of each cycle (1 cycle=28 days) while on treatment and for 30 days after the end of treatment
Description: Late adverse events (defined as any adverse events occur prior to diagnosis of progression/relapse and has not been previously reported) are collected via the long-term follow up forms at each follow-up visit.
Groups:
- MG 706+Octreotide: AMG 706 was administered on a flat scale of mg/day and not by weight or body surface area (BSA). AMG 706 was provided as a 25 mg tablet; the daily dose was 125 mg administered as five 25 mg tablets in the AM. AMG 706 was taken daily without breaks in treatment. Each cycle was defined as 28 days. AMG 706 was started within 7 working days of registration, given on the same day as the octreotide-LAR.
Arm/Group | MG 706+Octreotide
Serious Adverse Events (participants affected / at risk) | 26/45
Other Adverse Events (participants affected / at risk) | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MG 706+Octreotide (N=45)
Anemia (Blood and lymphatic system disorders) | 2
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Electrocardiogram QT corrected interval (Investigations) | 1
Hypertension (Vascular disorders) | 12
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 6
Weight loss (Investigations) | 1
INR increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 5
Urinary tract infection (Infections and infestations) | 1
Infections and infestations - blood (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Lipase increased (Investigations) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Ataxia (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MG 706+Octreotide (N=45)
Anemia (Blood and lymphatic system disorders) | 11
White blood cell decreased (Investigations) | 11
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 13
Hypertension (Vascular disorders) | 26
Hypotension (Vascular disorders) | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 7
Fatigue (General disorders) | 29
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Weight loss (Investigations) | 21
Anorexia (Metabolism and nutrition disorders) | 15
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 23
Abdominal distension (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 9
Edema limbs (General disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Alkaline phosphatase increased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less